CLINICAL TRIAL: NCT02565212
Title: Istanbul Gaziosmanpasa Taksim Research and Training Hospital,
Brief Title: Comparison of the Effects of Nasal Steroids and Montelukast on Olfactory Functions in Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, dalgic abdullah, Istanbul Gaziosmanpasa Taksim Research and Training Hospital,, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55
Record Dates: First submitted 2015-06-15; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Allergic Rhinitis
Keywords: Montelukast; Sniffin' Sticks test; allergic rhinitis; mometasone furoate
MeSH Terms: conditions — Rhinitis, Allergic | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- GROUP 1 (Experimental): montelukast sodium and mometasone
  Interventions: Drug: Montelukast,mometazon froat
- Group 2 (Active Comparator): montelukast
  Interventions: Drug: Montelukast,mometazon froat
- Group 3 (Active Comparator): mometasone furoate
  Interventions: Drug: Montelukast,mometazon froat

INTERVENTIONS:
Drug: Montelukast,mometazon froat

SUMMARY:
The investigators aimed to evaluate by the Sniffin' Sticks test the effects on olfactory functions of nasal steroids and leukotriene antagonists used for allergic rhinitis.Thirty patients with seasonal were included in this study. Patients were randomly divided into three groups of 10 patients; group 1 received montelukast sodium and mometasone furoate therapy, group 2 received only montelukast, and group 3 only mometasone furoate. Patients' olfactory functions were determined using the Sniffin' Sticks olfactory test before and after a month treatments.

Threshold, discrimination, identification, and TDI values were not significantly different among the groups before treatment. For Group 1 and Group 3 patients, there were statistically significant differences in threshold, discrimination, identification, and TDI values before and after treatment (p < 0.05) (Wilcoxon signed ranks analysis) For Group 2 patients, the before and after treatment values of threshold, discrimination, identification, and TDI showed no significant differences (p > 0.05). According to the findings of our study, MF is superior to montelukast in improving olfactory function. Although montelukast has been shown to be effective against AR symptoms, its effect on olfactory function was not demonstrated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Positive skin test to grass and/or tree pollens in patients with clinical history of seasonal AR for at least 1 year

Exclusion Criteria:

* Patients who had received drug treatment or immunotherapy before the study were excluded.
* Patients with asthma, deviated nasal septum, history of nasal operation, turbinate hypertrophy, nasal polyposis or chronic nasal disorders, pregnancy, or upper airway infections were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of nasal steroids and montelukast on olfactory functions in patients with allergic rhinitis | 1 month
  Sniff'in and Snick test (olfactory Test)